CLINICAL TRIAL: NCT02567643
Title: Stereotactic Radiosurgery for Multiple (5+) CNS Metastases
Brief Title: Stereotactic Radiosurgery (SRS) for Multiple CNS Mets
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-032
Record Dates: First submitted 2014-04-03; First posted 2015-10-05 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Cancer; Brain Metastases
Keywords: Brain; CNS; Metastases
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Radiosurgery (Experimental)
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery
  Other Names: Gamma Knife; Cyber Knife; SRS

SUMMARY:
This study is designed to determine outcome for patients with 5 or more central nervous system (CNS) metastatic lesions treated with stereotactic radiosurgery (SRS).

ELIGIBILITY:
Inclusion Criteria:

* CNS metastatic disease with 5 to 25 CNS mets that require treatment (note that previous SRS, WBRT, and resection for previous CNS mets is allowed. At time of protocol treatment, patient must have 5 or more new or progressing CNS mets that require treatment, this includes new lesions not before seen or progression of previous lesions.). While definition of new lesions is fairly straightforward, the definition of progression of old lesion is at the discretion of the treating team but it is recommended that progression be defined by a multidisciplinary team (radiation oncologist, neurosurgeon, neuro-radiologist). Note that treatment of tumor bed does not count as treatment of an active lesion.

For example,

* Patient with 10 lesions in 2010 who had whole brain radiation and now has 2 new lesions and progression of 3 previously noted lesions would be eligible
* Patient with 31 lesions in 2010 who had whole brain radiation and now has 26 stable lesions and progression of 5 lesions is eligible. Although the patient has more than 25 lesions the majority are stable and do not require treatment.
* Patient with 6 brain lesions has surgical resection of one lesion is eligible. Patient will require treatment for 5 lesions. Patient can also have treatment of surgical tumor bed but this does not count towards 5 lesions required for eligibility.
* All lesions < 4 cm in greatest dimension
* Able to have an MRI with contrast
* MRI within 6 weeks (MRI for eligibility can be done without contrast but planning MRI for radiosurgery will have contrast).
* Patients of child-bearing age must agree to contraception until radiosurgery has been completed.
* Patients able to undergo radiosurgery. Gamma knife radiosurgery is preferred for this protocol but cyberknife can also be used at the discretion of treating physicians.
* Karnofsky Performance Scale (KPS) 50 or better
* Eligible primaries:

  * Lung (NSCLC)
  * Lung (SCLC) that have had previous whole brain radiation
  * GI
  * Head and Neck
  * Gyn
  * Prostate
  * Breast
  * Kidney
  * Melanoma
  * Sarcoma

Exclusion Criteria:

* Less than 5 CNS lesions (can have had previously treated lesions by either surgery or SRS, but at time of protocol SRS must have 5 or more untreated lesions).
* More than 25 CNS lesions that require treatment (note that the patient can have had previous metastatic lesions, but at the time of enrollment cannot have more than 25 new lesions).

For example:

Patient with 12 brain lesions has whole brain radiation in 2010, on follow-up has progression of 3 lesions is not eligible since less than 5 lesions require treatment.

Patient with 5 brain lesions has surgical resection of one lesions, patient is not eligible since has less than 5 lesions that require treatment.

* Ineligible primaries Lymphoma Lung (SCLC) that have not had previous whole brain radiation Primary CNS tumors Leptomeningeal disease in CNS
* Must not have any chemotherapy or targeted therapy within 24 hours prior to SRS
* Patients unable to have an MRI (secondary for example to metal hardware)
* Patients unable to have MRI contrast (secondary for example to poor renal function).
* CNS lesion > 4 cm in any dimension
* KPS 40 or less
* Serious or other life threatening illness as determined by the treating physician

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | 6 months
Distant CNS free survival (new lesions in CNS) | 6 months

SECONDARY OUTCOMES:
Quality of life (as determined by FACT-Br) | 6 months
Local control (For CNS, local control refers to treated lesions) | 6 months
Timing and need for salvage therapy (whole brain radiation or repeat whole brain radiation) | 6 months
Median dose to whole brain with SRS | 6 months
Neurocognitive testing (Montreal Cognitive Assessment) | 6 months
Adverse Events for Safety and Tolerability of treatment | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center at Cooper, Camden, New Jersey, United States